CLINICAL TRIAL: NCT02337699
Title: DORSAL ROOT GANGLION STIMULATION AS TREATMENT FOR POSTSURGICAL GROIN PAIN (GASPA Study)
Brief Title: Dorsal Root Ganglion Stimulation as Treatment for Post-surgical Groin Pain
Acronym: GASPA
Status: Terminated | Type: Observational
Why Stopped: The Principal investigator retired without replacement. Only one patient was enrolled and completed the entire study without adverse events.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 25-SMI-2014
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Post Surgical Groin Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated Subjects: All subjects recruited into the main study treated with the Axium neurostimulator
  Interventions: Device: Implantation with the commercially available Axium neurostimulator
- QST Group: A sub-set of the main study group who also consent to take part in the Quantitative Sensory Testing based feasibility study
  Interventions: Device: Implantation with the commercially available Axium neurostimulator; Procedure: QST Testing

INTERVENTIONS:
Device: Implantation with the commercially available Axium neurostimulator
Procedure: QST Testing
  Groups: QST Group

SUMMARY:
25-SMI-2014 is a post market observational, questionnaire based study to assess the effectiveness of the Axium neurostimulator as a treatment for chronic post surgical groin pain. Within is also a nested feasibility study to assess the clinical utility of a Quantitive Sensory Testing (QST) protocol in the management of the described study group.

ELIGIBILITY:
Main Study

Inclusion Criteria:

1. Male
2. Age between >18 and <65 years
3. Unilateral post surgical groin pain for >6 months
4. Pain localized to the region defined by the anterior superior iliac spine (ASIS), the pubic tubercle, and the groin-gluteal-greater trochanter triangles (3G) point,
5. Pain has no surgical indication
6. Subjects meet the criteria for SCS implantation as set out in the Dutch Neuromodulation Society Guideline
7. Pain characterized by neuropathy and/or allodynia
8. Average daily baseline pain intensity baseline VAS greater than or equal to 50 mm on a 100mm VAS scale
9. Patient willing and able to give informed consent and to participate in observational study

Exclusion Criteria:

1. Inability to speak/read Dutch
2. Bilateral and/or recurrent hernia.
3. Radiofrequency or injection therapy at or close to a target DRG in the 90 days prior to enrolment
4. Current illicit drug use and/or alcohol dependence
5. Active infection, or conditions or indwelling devices that pose an increased risk of infection
6. Active implantable device including implantable cardiac defibrillator, pacemaker, spinal cord stimulator or intrathecal drug pump
7. Participation in another clinical study during the study period.
8. Any other disorder, condition, or circumstance that, in the opinion of the principal investigator, represents a risk to successful completion of all study activities.

Additional Criteria for nested feasibility study

Additional Inclusion Criteria

1. Participation in the observational study
2. Sign off for sub-study on patient informed consent

Additional Exclusion Criteria

1. For sub-study participation only: pain conditions [aside from the post surgical groin pain to be treated], extensive scar tissue, skin conditions, or sensorimotor abnormalities in the areas for QST assessments: the painful groin, the contralateral groin, the ipsilateral arm, and the contralateral hand

Ages: 18 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Chronic Post Surgical Groin Pain Patients
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Main Study: Pain Relief - Assessed be Change in Pain Intensity from Pre-Treatment Baseline | Post implantation at; 1, 3 and 6 months
Feasibility Study: To determine subject acceptance of the described QST methodology and protocol; assessed using a 5 point Likert scale | Baseline then Post implantation at; 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius Ziekenhuis, Nieuwegein, Netherlands